CLINICAL TRIAL: NCT07318844
Title: Stroke Volume at Rest and During Exercise in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ronan Berg, Professor, MD DMSc, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-25024676
Record Dates: First submitted 2025-08-31; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: stroke volume; test-retest; Acute exercise
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise bout (Experimental): A cardiopulmonary exercise test (CPET), during which stroke volume and heart rate are continuously measured
  Interventions: Other: Cardiopulmonary exercise test

INTERVENTIONS:
Other: Cardiopulmonary exercise test — The two study days are identical, and consist of stroke volume, heart rate and non-invasive blood pressure measurements during upright rest, in the supine position, and during incremental exercise (CPET).

SUMMARY:
Background Changes in cardiac output, driven by increased heart rate and stroke volume, are crucial for oxygen delivery during acute exercise and influence maximal oxygen uptake (VO₂max). Thoracic electrical bioimpedance provides a non-invasive alternative to traditional invasive methods by estimating stroke volume through impedance changes during ventricular filling and emptying. However, its test-retest reliability remains uncertain, requiring further investigation for use in acute and long-term training assessments.

Methods Inclusion: 12 healthy individuals (six males, six females) Exclusion: Known ischaemic heart disease, known heart failure, symptoms of disease within 2 weeks prior to the study, known malignant disease, claudication, pregnancy, unstable cardiac arrhythmic disease, renal or liver dysfunction, known chronic lung disease Design: Test-retest study of thoracic electrical bioimpedance-based stroke volume

Intervention: Acute exercise bout on a bicycle ergometer Statistical design: Rest-to-exercise changes, as well as between-day smallest real difference, coefficient of variation and intraclass correlation coefficient Sample size: Since this is a pilot study, the sample size is set at 12 in accordance with current recommendations.

Perspective The results are relevant for designing future studies in which stroke volume is measured and compared in response to various interventions at rest and during exercise.

ELIGIBILITY:
Inclusion criteria

* Men and women
* 18-70 years

Exclusion criteria

* Known chronic lung disease
* Known ischaemic heart disease
* Known heart failure
* Symptoms of disease within 2 weeks prior to the study
* Known malignant disease
* Claudication
* Pregnancy
* Unstable cardiac arrhythmic disease
* Renal or liver dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Between-day smallest real difference (SRD) for stroke volume during upright rest | 2-10 days
Between-day coefficient of variance (CV) for for stroke volume during upright rest | 2-10 days

SECONDARY OUTCOMES:
Between-day smallest real difference (SRD) for stroke volume during supine rest | 2-10 days
Between-day coefficient of variance (CV) for stroke volume during supine rest | 2-10 days
Between-day SRD for stroke volume at 60% of maximal workload (Wmax) during CPET | 2-10 days
Between-day CV for stroke volume at 60% of Wmax during CPET | 2-10 days

OTHER OUTCOMES:
Between-day SRD for stroke volume at 40% of Wmax during CPET | 2-10 days
Between-day CV for stroke volume at 40% of Wmax during CPET | 2-10 days
Between-day SRD for stroke volume at 80% of Wmax during CPET | 2-10 days
Between-day CV for stroke volume at 80% of Wmax during CPET | 2-10 days
Between-day SRD for stroke volume at Wmax during CPET | 2-10 days
Between-day CV for stroke volume at Wmax during CPET | 2-10 days
Between-day intraclass correlation coefficient (ICC) for stroke volume during upright rest | 2-10 days
Between-day ICC for stroke volume during supine rest | 2-10 days
Between-day ICC for stroke volume at 60% of Wmax during CPET | 2-10 days
Between-day ICC for stroke volume at 40% of Wmax during CPET | 2-10 days
Between-day ICC for stroke volume at 80% of Wmax during CPET | 2-10 days
Between-day ICC for stroke volume at Wmax during CPET | 2-10 days
Between-day SRD for cardiac output (measured as the product of stroke volume and heart rate) during upright rest | 2-10 days
Between-day CV for for cardiac output during upright rest | 2-10 days
Between-day ICC for for cardiac output during upright rest | 2-10 days
Between-day SRD for cardiac output during supine rest | 2-10 days
Between-day CV for for cardiac output during supine rest | 2-10 days
Between-day ICC for for cardiac output during supine rest | 2-10 days
Between-day SRD for cardiac output at 60% of Wmax during CPET | 2-10 days
Between-day CV for cardiac output at 60% of Wmax during CPET | 2-10 days
Between-day ICC for cardiac output at 60% of Wmax during CPET | 2-10 days
Between-day SRD for cardiac output at 40% of Wmax during CPET | 2-10 days
Between-day CV for cardiac output at 40% of Wmax during CPET | 2-10 days
Between-day ICC for cardiac output at 40% of Wmax during CPET | 2-10 days
Between-day SRD for cardiac output at 80% of Wmax during CPET | 2-10 days
Between-day CV for cardiac output at 80% of Wmax during CPET | 2-10 days
Between-day ICC for cardiac output at 80% of Wmax during CPET | 2-10 days
Between-day SRD for cardiac output at Wmax during CPET | 2-10 days
Between-day CV for cardiac output at Wmax during CPET | 2-10 days
Between-day ICC for cardiac output at Wmax during CPET | 2-10 days
Between-day SRD for heart rate (measured with the CPET equipment) during upright rest | 2-10 days
Between-day CV for for heart rate during upright rest | 2-10 days
Between-day ICC for for heart rate during upright rest | 2-10 days
Between-day SRD for heart rate during supine rest | 2-10 days
Between-day CV for for heart rate during supine rest | 2-10 days
Between-day ICC for for heart rate during supine rest | 2-10 days
Between-day SRD for heart rate at 60% of Wmax during CPET | 2-10 days
Between-day CV for heart rate at 60% of Wmax during CPET | 2-10 days
Between-day ICC for heart rate at 60% of Wmax during CPET | 2-10 days
Between-day SRD for heart rate at 40% of Wmax during CPET | 2-10 days
Between-day CV for heart rate at 40% of Wmax during CPET | 2-10 days
Between-day ICC for heart rate at 40% of Wmax during CPET | 2-10 days
Between-day SRD for heart rate at 80% of Wmax during CPET | 2-10 days
Between-day CV for heart rate at 80% of Wmax during CPET | 2-10 days
Between-day ICC for heart rate at 80% of Wmax during CPET | 2-10 days
Between-day SRD for heart rate at Wmax during CPET | 2-10 days
Between-day CV for heart rate at Wmax during CPET | 2-10 days
Between-day ICC for heart rate at Wmax during CPET | 2-10 days
Uright-to supine changes in stroke volume, heart-rate and cardiac output and arterial blood pressure at rest | 2-10 days
Changes in stroke volume from upright rest to exercise at 40%, 60%, 80% and 100% of Wmax. | 2-10 days
Changes in cardiac output from upright rest to exercise at 40%, 60%, 80% and 100% of Wmax. | 2-10 days
Changes in arterial blood pressure from upright rest to exercise at 40%, 60%, 80% and 100% of Wmax. | 2-10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Trygfondens Center for Aktiv Sundhed, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No